CLINICAL TRIAL: NCT06660303
Title: Preoperative Patient Education for Enhanced Recovery After Colon and Rectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elsayed Zaky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Preoperative Patient Education
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Colo-rectal Cancer
Keywords: Preoperative Education; Nursing Intervention; Enhanced Recovery After Surgery (ERAS)
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Patients who will receive comprehensive preoperative education tailored to their upcoming colorectal surgery. This education covers what to expect during the surgical process, postoperative care, pain management strategies, and guidelines to aid faster recovery.
  Interventions: Behavioral: Comprehensive Preoperative Education for Enhanced Recovery in Colorectal Surgery
- Control Group (Active Comparator): Participants which will receive routine hospital care. This means that participants in this group will go through the standard preoperative and postoperative procedures typically provided at the hospital without any additional specialized preoperative education or targeted nursing instructions
  Interventions: Other: Routine hospital care

INTERVENTIONS:
Behavioral: Comprehensive Preoperative Education for Enhanced Recovery in Colorectal Surgery — The intervention in this study involves preoperative patient education aimed at improving outcomes for individuals undergoing colorectal surgery. Patients in the study group will receive targeted educational sessions that focus on setting expectations, managing anxiety, understanding pain control, and preparing for the surgical process as part of the Enhanced Recovery After Surgery (ERAS) protocol. This educational approach is designed to empower patients, reduce anxiety, enhance satisfaction, and potentially improve post-surgical recovery compared to those receiving routine hospital care.
  Arms: Study group
Other: Routine hospital care — The control group, designated as Group II, will receive standard hospital care, encompassing the usual preoperative and postoperative procedures provided by the hospital. This includes typical preparation and recovery guidelines without any added specialized preoperative education or targeted nursing instructions. This routine hospital care serves as a baseline, allowing for a direct comparison of outcomes against the intervention group, which will receive comprehensive preoperative education aimed at enhancing recovery and improving surgical outcomes.
  Arms: Control Group

SUMMARY:
The aim of this experimental study is to evaluate whether **preoperative patient education can improve outcomes for individuals undergoing colorectal surgery. This study will focus on adult male and female patients with colon cancer scheduled for colorectal surgery through colonoscopy, excluding those undergoing open surgery.

The primary questions this study seeks to answer are:

* Do patients who receive preoperative education experience significantly lower levels of preoperative anxiety compared to those receiving routine hospital care?
* Do patients receiving nursing instructions report significantly lower levels of oral pain postoperatively compared to those who do not?
* Does preoperative education lead to higher levels of patient satisfaction compared to standard care?

Researchers will compare a study group that receives preoperative education to a control group receiving routine hospital care to determine the effectiveness of the intervention.

Participants will be asked to:

* Complete a demographic and medical history questionnaire.
* Utilize the Pain Numeric Rating Scale (NRS-11) to self-report pain levels.
* Participate in assessments using the Amsterdam Preoperative Anxiety and Information Scale (APAIS)**.
* Complete a satisfaction survey using the Colorectal Surgical Patient's Satisfaction Tool after surgery.

The study aims to assess the impact of preoperative education on anxiety, pain management, and overall patient satisfaction.

DETAILED DESCRIPTION:
Patient education and engagement are fundamental components of modern integrated colorectal care pathways. Surgeons and nurses play a crucial role in providing comprehensive education about what patients can expect during both the preoperative and postoperative phases of surgery. Setting clear expectations early-especially regarding the anticipated discharge date-significantly influences the postoperative recovery journey.

Enhanced Recovery After Surgery (ERAS) is an evidence-based, patient-focused strategy aimed at optimizing surgical outcomes by streamlining the recovery process. Initially designed for colorectal procedures, ERAS protocols have now been adapted for various surgical disciplines, with many of its principles safely applicable to most perioperative patients. The primary objective of ERAS is to minimize the physical and emotional strain of surgery, facilitating quicker recovery, reducing complications, and decreasing the length of hospital stays.

While much of the research on the ERAS program has traditionally centered on the surgeon's role, the multidisciplinary nature of patient care has brought increased recognition to the nurse's contribution. Nursing professionals are now acknowledged as vital components of the ERAS framework, playing a key role in ensuring the program's success.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients with colon cancer undergoing colorectal surgery via colonoscope.

Exclusion Criteria:

* patients with open surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Pain Rating Scale | 1 week
  pain Numeric Rating Scale (NRS-11) is 10-point scale for patient self-reporting of pain. It is for adults as 0 indicates no pain, 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain.

SECONDARY OUTCOMES:
Amsterdam preoperative anxiety and information scale (APAIS) | 1 week
  is scale consists of four items (questions 1, 2, 4, 5), each of which could be scored from 1 to 5. The score of the anxiety scale is the sum of these four questions, with a scoring range from 4 to 20.it is developed by Moerman, van Dam, Muller & Oosting. (1996). Reliability was 0.74.

OTHER OUTCOMES:
Colorectal Surgical Patient's Satisfaction tool | 1 week
  Likert scale ranging from 1 to 3; a score(1) dissatisfied, (2) neutral, (3) satisfied. The total score value ranged between 15 - 45. The higher the score the higher the patient's satisfaction level. This tool was adopted from Salisbury et al., (2005). It was translated to Arabic language and tested for validity and reliability by Abd El-Aziz, (2011). Its internal consistency reliability was (r = 0.840).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculy of Nursing Cairo University, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Dipokromo, A., Sherman, D. W., & Lago Sr, C. (2022). Preoperative Education Regarding the Enhanced Recovery After Surgery (ERAS) Guideline for colorectal Surgical Patients: A Quality Improvement Project.
- [Background] Carrilho, M. P. G., Pontífice-Sousa, P., & Marques, R. M. D. (2021). ERAS® Program-Nursing care for patients undergoing colorectal surgery. Acta Paulista de Enfermagem, 34, eAPE002105.
- [Background] Abd El-Aziz E. The Effect of the Application of Clinical Pathway on Postoperative Outcomes of Patients Undergoing Percutaneous Nephrolithotomy. Alexandria University, Faculty of Nursing: Unpublished DSN dissertation. 2011.